CLINICAL TRIAL: NCT03493646
Title: Evaluating in Vivo AZA Incorporation in Mononuclear Cells Following Vidaza or CC486
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01-AZA; VZ-CL-MDSAML-PI-13085 (Other: Kirby Institute)
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic Syndrome; MDS; Acute Myeloid Leukemia; AML; Chronic Myelomonocytic Leukemia; CMML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; cc-486

STUDY DESIGN:
Intervention Model Description: Phase II open label multicentre study. All participants will commence with Vidaza for 6 cycles, followed by 6 cycles of CC 486 regardless of response to Vidaza
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azacitidine (Active Comparator): 6 cycles of azacitidine (28 day cycle)
  Interventions: Drug: Azacitidine
- CC 486 (Experimental): 6 cycles CC 486 (28 day cycle)
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: Azacitidine — 75mg/m2 per day for 7 days of each 28 day cycle. Cycles 1-6
  Other Names: Vidaza
  Arms: Azacitidine
Drug: CC-486 — 100 mg BID for the first 21 days of each 28-day treatment cycle (cycles 7-8). The dose should be increased from cycle 9 onwards to 150mg BID for the first 21 days of each 28-day treatment cycle (cycles 9-12) in the absence of Grade 3 or 4 AE. If 2 or more cycles are tolerated at this dose, further increments are permitted for patients with Stable Disease or if clinically indicated in consultation with the coordinating investigator as per the study dose modification schedule.
  Other Names: Oral azacitidine
  Arms: CC 486

SUMMARY:
Myelodysplastic Syndrome (MDS) is a group of blood disorders where the bone marrow does not produce enough mature red blood cells, white blood cells and platelets. In a healthy person, the bone marrow makes blood stem cells (immature cells, also called 'blasts') that become mature blood cells over time. In people with MDS, this process is affected and immature blood cells in the bone marrow do not mature fully to become healthy blood cells. This causes a lack of healthy blood cells that can function properly. With fewer healthy blood cells, infection, anaemia, or easy bleeding may occur. MDS can progress to acute myeloid leukaemia in 25-30% of patients, and if untreated it can be rapidly fatal.

The purpose of this study is to evaluate the standard treatment, azacitidine (Vidaza) given as an injection under the skin compared to the same medication (called CC-486) taken as a tablet by mouth. Vidaza is approved by the Australian Therapeutics Goods Administration (TGA) as standard treatment for MDS. CC-486 is an experimental treatment. This means it is not an approved treatment for MDS in Australia. CC-486 is being developed to increase convenience and make it easier for patients to continue their treatment. So far it has been given to over 870 patients in studies across the world. The treatment in the injection and the tablet is the same. Studies like this one are being done to ensure the tablet works in the same way as the standard injected treatment.

Vidaza is given by subcutaneous injection (ie under the skin) over an hour for 7 days every 4 weeks for as long as it continues to work. All study participants will receive active treatment (there is no placebo), and all participants will receive the standard injection for six treatment cycles followed by the new tablet medication taken once daily for 21 days every 4 weeks. This allows the researchers to compare the two ways of giving the medicine.

DETAILED DESCRIPTION:
MDS is an insidious and largely incurable haematological malignancy that increasingly impacts on the well-being of our ageing population, and one for which there has been no significant therapeutic advance since the introduction of injectable AZA (Vidaza®) over a decade ago.

Furthermore, the basis for the effectiveness of Vidaza® or lack thereof is not known and attempts at identifying genes that are reactivated and induce HSC differentiation have generally been unrewarding. It is also unclear whether these drugs work by inducing cellular differentiation or triggering apoptosis of the abnormal clone by activating permissive gene transcription. Recently developed assays permit genome-wide mutation analysis and assessment of gene expression and methylation at gene regulatory regions. Combined with functional studies, these assays are powerful tools that could help identify why some patients respond and others don't and why patients relapse after initial response. They can also help provide molecular insights into specific genes or pathways that could be manipulated to overcome primary or secondary drug resistance to AZA.

Following the evaluation CC-486 safety in Phase 1 studies, a Phase 2, international, multicentre, randomized, open-label, parallel group study was launched and is currently recruiting to evaluate the efficacy and safety of CC-486 alone and in combination with durvalumab in participants with MDS who fail to achieve objective response to treatment with Vidaza®. However, at present there is no objective method of correlating clinical or molecular response with actual drug incorporation due to the lack of a robust assay to measure AZA incorporation in vivo.

This gap has now been filled by the recent development of a liquid chromatography-mass spectrometry (LC-MS) based assay that is effective in measuring AZA pharmacokinetics in vivo; "AZA-MS: a novel mass spectrometry method to determine the intracellular pharmacokinetics of AZA therapy in vivo" (Unnikrishnan et al Leukemia 2017) and we will for the first time be able to directly compare Vidaza® incorporation with CC486 incorporation in the same patient and measuring clinical and molecular response after six cycles of the former followed by six cycles of the latter. The primary objective of the trial is to determine whether there is greater AZA incorporation in DNA in blood progenitors following 21 days of CC486 than there is with 7 days of Vidaza® in a 28- day treatment cycle and whether incorporation is associated with greater clinical and/or molecular response.

The secondary objectives of the trial are based on outcomes from a compassionate access program conducted in NSW, Australia from 2008-09. MDS, MDS/AML and CMML patients who respond to Vidaza® were found to have a greater fraction of hematopoietic progenitor cells (HPCs) progressing through the cell cycle than patients who fail to respond to AZA (Unnikrishnan et al 2017). What is not known is whether increased replication is associated with increased AZA incorporation. The availability of an assay (AZA-MS) to measure AZA incorporation, and the ability to measure the fraction of replicative HPCs, forms the basis of the secondary objectives of this study.

When applying the AZA-MS assay to samples collected from the compassionate access program, we also noted that AZA non-responders either do not incorporate AZA derivatives in DNA following Vidaza® or do incorporate AZA to levels comparable to that of responders yet still fail to respond (Unnikrishnan et al Leukemia 2017). Mechanisms of pharmacologically overcoming resistance would be quite different in the two instances. Longitudinal measurements of derivative AZA incorporation in DNA can now be combined with assays to evaluate whether patients who do not respond despite adequate drug uptake fail to activate downstream processes such as interferon/immune pathway activation or display check-point inhibition. This study will provide data to support individualised alternatives to optimise future AZA therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age.
2. Documented diagnosis of

   1. Myelodysplastic syndrome classified as intermediate-2 or high risk according to the IPSS, or
   2. AML with 20-30% marrow blasts and multi-lineage dysplasia, according to WHO classification, or
   3. CMML with 10-29% marrow blasts without myeloproliferative disorder according to WHO classification, or Confirmation will be from either the BMA performed at screening or a standard of care BMA if performed up to 6 weeks before cycle 1 day 1.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
4. Females of childbearing potential (FCBP) may participate, providing they meet the following conditions:

   1. Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; true abstinence; or vasectomized partner) throughout the study, and for 90 days following the last dose of investigational product (IP); and
   2. Have a negative serum pregnancy test at screening
5. Male participants with a female partner of childbearing potential must agree to use at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 90 days following the last dose of Investigational Product.
6. Understand and voluntarily sign an informed consent document prior to any study- related assessments or procedures conducted.

Exclusion Criteria:

1. Acute myeloid leukemia (AML) - ≥ 30% blasts in bone marrow according to WHO classification. Participants known to have ≥ 30% blasts are not eligible for inclusion in this study. Recognizing limitations of blast cell quantitation, this protocol will allow participants with pre-enrollment (screening/baseline) bone marrow blast counts up to 33% to be considered for inclusion subject to discussion with the Coordinating PI prior to enrollment.
2. Prior allogeneic or autologous stem cell transplant.
3. Prior exposure to a hypomethylating agent.
4. Use of any of the following within 28 days prior to cycle 1, day 1:

   1. thrombopoiesis-stimulating agents ([TSAs]; eg, Romiplostim, Eltrombopag, Interleukin-11)
   2. ESAs (Erythropoiesis stimulating agent) and other RBC hematopoietic growth factors (eg, interleukin-3)
   3. Hydroxyurea
   4. Any other investigational product from another clinical trial
5. Concurrent use of corticosteroids unless the participant is on a stable or decreasing dose for ≥ 1 week prior to enrollment for medical conditions other than MDS.
6. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the IP and/or predispose the participant to an increased risk of gastrointestinal toxicity.
7. Prior history of malignancies, other than MDS, unless the participant has been free of the disease for ≥ 3 years. However, participants with the following history/concurrent conditions are allowed:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
8. Significant active cardiac disease within the previous 6 months, including:

   1. New York Heart Association (NYHA) class IV congestive heart failure
   2. Unstable angina or angina requiring surgical or medical intervention; and/or
   3. Myocardial infarction
9. Active systemic infection including:

   1. Ongoing signs/symptoms related to the infection without improvement despite appropriate anti-infectives
   2. Active Hepatitis B infection
   3. Subjects with Human Immunodeficiency Virus (HIV) or Hepatitis C infection will be considered individually by the coordinating principal investigator:

   i) Those with HIV will generally be eligible if receiving antiretroviral therapy, HIV VL is suppressed <50 copies/mL and CD4≥350 cells/mm3. ii) Those with HCV will generally be eligible if there is no evidence of clinical hepatic dysfunction or other systemic manifestations of HCV disease and the hepatic parameters below are met. Consideration should be given to curative HCV therapy prior to enrollment in consultation with HCV clinician, if possible.
10. Any of the following laboratory abnormalities:

    1. Serum AST/SGOT or ALT/SGPT > 2.5 x ULN
    2. Serum total bilirubin > 1.5 x ULN. Higher levels are acceptable if these can be attributed to active RBC precursor destruction within the bone marrow (ie, ineffective erythropoiesis).
    3. Evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Direct Antiglobulin Test or over 50% of indirect bilirubin
    4. Serum creatinine > 2.5 x ULN
    5. Absolute white blood cell count ≥ 20 x 109/L
11. Known or suspected hypersensitivity to azacitidine, mannitol, its constituents, or to any other humanized monoclonal antibody.
12. Pregnant or breast-feeding females.
13. Clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia.
14. Any condition not already outlined above which, in the opinion of the clinical investigator, would place the subject at risk if they participated or would jeopardise adherence or follow up or confound the ability to interpret study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
DNA incorporation of Vidaza® compared to CC-486 | At the end of cycle 6 (cycles 1-6 inclusive) compared with cycles 7-12 (cycles 7-12 inclusive). Each cycle is 28 days
  DNA incorporation of Vidaza® compared to CC-486 as measured by the area under the curve (AUC) during the first 6 cycles compared to the area under the curve from cycles 7 to 12.

SECONDARY OUTCOMES:
DNA incorporation in bone marrow mononuclear cells | At the end of cycle 6 compared to cycle 7. Each cycle is 28 days
  DNA incorporation in bone marrow mononuclear cells following Vidaza® compared to CC-486 as measured by the area under the curve (AUC) in cycle 6 compared to the AUC in cycle 7
DNA AZA derivative uptake | end of Cycle 6 and 12
  DNA AZA derivative uptake (measured by AUC) between responders and non-responders who are classified as having AZA uptake
Proportion of cells undergoing the cell cycle | end of Cycle 6 and 12. Each cycle is 28 days
  Proportion of cells undergoing the cell cycle for non-responders with AZA uptake vs non-responders without AZA uptake
Inflammatory markers, as measured by AUC, between responders and non- | end of Cycle 6 and 12. Each cycle is 28 days
  Inflammatory markers, as measured by AUC, between responders and non-responders who are classified as having AZA uptake

CONTACTS AND LOCATIONS:
Overall Officials: John Pimanda, MD, Principal Investigator — University of New South Wales
Locations (11):
- Australia (11):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Gosford and Wyong Hospitals, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - St Vincent's hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided